CLINICAL TRIAL: NCT00929396
Title: A Safety and Immunogenicity Phase 1 Trial With an Adjuvanted TB Subunit Vaccine (Ag85B-ESAT-6 + IC31)Administered in PPD Positive Volunteers at 0 and 2 Months
Brief Title: A Safety and Immunogenicity Trial With an Adjuvanted Tuberculosis (TB) Subunit Vaccine in Purified Protein Derivative (PPD) Positive Volunteers
Acronym: THYB-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THYB-02
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Ag85B; ESAT-6; IC31
MeSH Terms: conditions — Tuberculosis | interventions — Adjuvants, Pharmaceutic; IC31 adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Latent TB infection group (Experimental): The latent TB group will receive two injections of 50 microgram antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a)two months apart.
  Interventions: Biological: 50 microg. antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a)
- BCG vaccinated group (Experimental): The BCG vaccinated group will receive two vaccinations of 50 microgram antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a)two months apart
  Interventions: Biological: 50 microg. antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a)

INTERVENTIONS:
Biological: 50 microg. antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a) — o,5 mL suspension for injection x 2 with 2 months interval
  Other Names: Antigen H1 + adjuvant IC31
  Arms: BCG vaccinated group
Biological: 50 microg. antigen + adjuvant (500 nmol KLK + 20 nmol ODN1a) — o,5 mL suspension for injection x 2 with 2 months interval
  Other Names: Antigen H1 + adjuvant IC31
  Arms: Latent TB infection group

SUMMARY:
The purpose of this study is to evaluate the safety profile of an adjuvanted TB subunit vaccine administered at 0 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 55 years old
* BCG group: Known to be BCG-vaccinated over 2 years before, PPD positive (range 6-15 mm or any documented value between 6-15 mm on medical file in the past), with no active, chronic or past TB disease as confirmed by chest X ray, negative QuantiFERON-TB Gold In Tube test and negative 6-day lymphocyte tests.
* Infection group: Known to be treated for latent TB, PPDpositive (equal or over 10 mm or documented equal or over 10 mm positive on medical file in the past), previously TB infected but with no active disease confirmed by chest X ray, may have received chemoprophylaxis but with no TB treatment/chemoprophylaxis within the preceding 2 years, positive QuantiFERON-TB Gold In Tube test and/or positive 6-day lymphocyte test.
* Healthy based on medical examination/history at the inclusion
* Signed informed consent
* Prepared to grant authorized persons access to the medical records
* The volunteer is likely to comply with instructions

Exclusion Criteria:

* Granulomatous disease (by chest X-ray)
* Vaccinated with live vaccine 3 months before first vaccination
* Administration of immune modulating drugs (steroids, immunosuppressive drugs or immunoglobulins) 3 months before the first vaccination
* HBV, HCV or HIV sero-positive
* Participation in other clinical trials
* Known hypersensitivity to any of the vaccine components
* Laboratory parameters outside of normal range judged by PI to be clinically relevant
* Pregnant women/planned pregnancy and/or breastfeeding within the trial period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Physical examination. Local adverse events.Systemic adverse events. Laboratory safety tests including urine safety tests. | From first vaccination until 8 months after the first vaccination

SECONDARY OUTCOMES:
Detection by ELISPOT of IFNgamma spot-forming cells in PBMCs. Detection by ELISA of IFNgamma production in supernatants of PBMC. Detection by ELISA of IgG antibodies in serum/plasma. Detection by Elisa of TNFalfa and IFNgamma in serum | From first vaccination until 8 months after first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jaap van Dissel, MD, Prof., Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, RC Leiden, Netherlands

REFERENCES:
- [Derived] van Dissel JT, Soonawala D, Joosten SA, Prins C, Arend SM, Bang P, Tingskov PN, Lingnau K, Nouta J, Hoff ST, Rosenkrands I, Kromann I, Ottenhoff TH, Doherty TM, Andersen P. Ag85B-ESAT-6 adjuvanted with IC31(R) promotes strong and long-lived Mycobacterium tuberculosis specific T cell responses in volunteers with previous BCG vaccination or tuberculosis infection. Vaccine. 2011 Mar 3;29(11):2100-9. doi: 10.1016/j.vaccine.2010.12.135. Epub 2011 Jan 20. PMID 21256189